CLINICAL TRIAL: NCT02982681
Title: COMPARATIVE EVALUATION OF BIOACTIVE GLASS PUTTY AND PLATELET RICH FIBRIN IN THE TREATMENT OF HUMAN PERIODONTAL INTRABONY DEFECTS- A CLINICAL AND RADIOGRAPHICAL STUDY"
Brief Title: Bioactive Glass and Platelet Rich Fibrin in Intrabony Defects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. D. Y. Patil Dental College & Hospital (Other)
Collaborators: Santosh University (Other)
Responsible Party: Principal Investigator, Santosh Martande, Assistant Professor, Dr. D. Y. Patil Dental College & Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUG/25/2015
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Periodontal Diseases; Bone Resorption
Keywords: Periodontal disease; Platelet rich fibrin
MeSH Terms: conditions — Periodontal Diseases; Bone Resorption | interventions — Bioglass

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platelet rich Fibrin (Experimental): The intrabony defects were treated with Full thickness mucoperiosteal flap was raised and thorough open flap debridement done under local anesthesia In the test site the graft was then carefully compacted from the base of the defect coronally. PRF membrane was placed in the test site secured with vicryl sutures.
  Interventions: Drug: Platelet rich fibrin
- Bioactive glass (Active Comparator): The intrabony defects were treated with Full thickness mucoperiosteal flap was raised and thorough open flap debridement done under local anesthesia and The control site were packed with the graft alone
  Interventions: Drug: Bioactive Glass

INTERVENTIONS:
Drug: Platelet rich fibrin — In the test site the graft was then carefully compacted from the base of the defect coronally. PRF membrane was placed in the test site
  Other Names: PRF
  Arms: Platelet rich Fibrin
Drug: Bioactive Glass — The control site were packed with the bioactive glass graft alone
  Other Names: Novabone
  Arms: Bioactive glass

SUMMARY:
Background: Platelet-rich fibrin (PRF) and bioactive glass putty has been shown to be effective in promoting reduction in probing depth, gain in clinical attachment, and defect fill in intrabony periodontal defects. The individual role played by bioactive glass putty in combination with PRF is yet to be elucidated.

AIM: To compare the clinical effectiveness of the combination of Plaltelet Rich Fibrin and Bioactive Glass Putty and Bioactive glass putty regenerative techniques for intrabony defects in humans.

Material and methods: Ten pairs of intrabony defects were surgically treated with PRF and Bioactive glass putty (Test group) on one side or bioactive glass putty (Control group) on other side. The primary outcomes of the study included changes in probing depth, attachment level and bone fill of Osseous defect. The clinical parameters were recorded at baseline, 3, 6, and 9 months. Radiographic assessment was done using standardized intra oral periapical radiographs. Comparisions were made within each group between baseline, 3 months, 6 months and 9 months using the ANOVA test followed by Bonferroni test.

DETAILED DESCRIPTION:
INTRODUCTION

Periodontitis is an infectious disease that causes destruction of the attachment apparatus.[1].The mainstay aim of periodontal treatment is the regeneration of the lost attachment apparatus of the teeth. Variety of treatment modalities are available for periodontal regenerative therapy including bone grafts, bone substitutes, Guided Tissue Regeneration, growth factors, application of tissue engineering or the combination of two or more of the above listed approaches. [2] Alloplasts, may be an effective alternative to allograft and xenografts as there is no risk of disease transmission and the supply is unlimited.[3] The Bioactive glass promotes osteogenesis by adsorption and concentrations of protein utilized by osteoblast to form a mineralized extracellular matrix. [4] The advantage of the putty form of bioactive glass is the glycerine and polyethylene glycol which makes the glass particle coherent and thus enhancing handling characteristics and minimal migration of graft particles from the defect site. [5] Histological evaluation of material has shown that the particulate tends to retard the down growth of epithelial tissue. [6,7,8,9] Growth factors play a pivotal role in periodontal regeneration. Platelet Rich Fibrin is believed to release polypeptide growth factors, such as transforming growth factors-ß, platelet derived growth factors, vascular endothelial growth factors and matrix glycoproteins (such as thrombospondin -1) into the surgical wound in a sustained fashion for at least 7 days as shown in vitro. [10] Thus, given the unique graft with osteoconductive, osteoinductive and osteostimulative properties and properties of autologous PRF, application of combination approach was attempted for the assessment of their additional benefits to the healing mechanisms and periodontal regeneration in intrabony defects.

Materials and methods Patient Selection This randomized control trial was carried out in the Department of Periodontics and Oral Implantology, Santosh Dental College and Hospital, Santosh University, Ghaziabad. Ten patients suffering chronic localized periodontitis aged between 20 -50 years (7 males and 3 females) with 10 pairs of contalateral intraosseous defects (n=20) comprised the study population. A total of 20 bone defects (10 pairs) were decided by the statisticion to be of statistical strength. Convenient sampling design was used for the enrolment of study patients. Ethical approval was taken from the institutional ethical committee The patients were explained in detail about the procedure and a written informed consent was taken. The intrabony defects were diagnosed clinically with moderate to deep periodontal pockets > or = 5mm and with clinical and radiographic evidence of vertical/angular osseous defects. [3] Patients with systemic diseases, on anticoagulants, those with habit of smoking and alcohol, with known history of allergy to graft material and who have undergone periodontal surgical treatment for chronic periodontitis within twelve months for the same defects were excluded from the study.

PRESURGICAL THERAPY Patients underwent phase I therapy. The selected defects were evaluated after 2 weeks, and persistent pockets > or = 5mm and patients with clinical radiographic evidence of angular osseous defects were scheduled for surgery.

Clinical Parameters :

Oral hygiene status was recorded using the gingival index of Loe & Sillness,[11];

with score 0 indicating absence of inflammation and score 3 indicating severe

inflammation and plaque index of Silness & Loe. [12]

Probing pocket depth and Clinical attachment level were recorded at baseline on the

day of surgery, 3, 6 and 9 months intervals using UNC-15 probe and customized

acrylic occlusal stents grooved in the area of defect to provide reproducible insertion

axis-

The following measurements were recorded with customized

acrylic stent:

* Fixed reference point (FRP) to the base of pocket (BP)
* Fixed reference point (FRP) to the cemento-enamel junction (CEJ)
* Fixed reference point (FRP) to the gingival margin (GM)

PPD and CAL were calculated from these probing measurements as:

* PPD = (FRP to BP) - (FRP to GM)
* CAL= (FRP to BP) - (FRP to CEJ)

Radiographic measurements: Standardized intra-oral periapical radiographs of the defects were taken using a paralleling technique.[13]

Amount of defect fill: Defects were measured from the fixed reference point (distance between the cemento-enamel junction to the radiographic base of the bone defect ) with the help of 1.1 mm grid and the following radiographic features were recorded on the day of surgery, 3, 6 and 9 months intervals.

ELIGIBILITY:
Inclusion Criteria:

* The intrabony defects were diagnosed clinically with moderate to deep periodontal pockets > or = 5mm and with clinical and radiographic evidence of vertical/angular osseous defects.

Exclusion Criteria:

* Patients with systemic diseases, on anticoagulants, those with habit of smoking and alcohol, with known history of allergy to graft material and who have undergone periodontal surgical treatment for chronic periodontitis within twelve months for the same defects were excluded from the study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Intrabony defect fill | baseline to 9 months
  change in intrabony defect fill from baseline to 9 months

SECONDARY OUTCOMES:
Probing depth | baseline to 9 months
  change in probing depth from baseline to 9 months
Clinical attachment level | baseline to 9 months
  change in Clinical attachment level from baseline to 9 months
Gingival Index | baseline to 9 months
  change in Gingival Index from baseline to 9 months

REFERENCES:
- [Background] Hall EE, Meffert RM, Hermann JS, Mellonig JT, Cochran DL. Comparison of bioactive glass to demineralized freeze-dried bone allograft in the treatment of intrabony defects around implants in the canine mandible. J Periodontol. 1999 May;70(5):526-35. doi: 10.1902/jop.1999.70.5.526. PMID 10368057
- [Background] Dohan Ehrenfest DM, de Peppo GM, Doglioli P, Sammartino G. Slow release of growth factors and thrombospondin-1 in Choukroun's platelet-rich fibrin (PRF): a gold standard to achieve for all surgical platelet concentrates technologies. Growth Factors. 2009 Feb;27(1):63-9. doi: 10.1080/08977190802636713. PMID 19089687